CLINICAL TRIAL: NCT01458262
Title: Observational Study on the Clinical Impact of Systemic and Cerebral Desaturation During Liver Transplantation and Hepatectomy
Brief Title: Observational Study on the Clinical Impact of Desaturation During Liver Surgery
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: CE10.192
Record Dates: First submitted 2011-09-22; First posted 2011-10-24 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Cerebral Desaturation
Keywords: cerebral oxymetry; systemic oxymetry; hepatic surgery; liver transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: systemic and cerebral oxymetry — oxymetry measurement using near infrared spectroscopy
  Other Names: oxymetry measurement using near infrared spectroscopy

SUMMARY:
The purpose of this study is to determine the clinical impact of cerebral and systemic desaturation during liver transplantation and resection on post-operative complications.

DETAILED DESCRIPTION:
This is an observational study. Cerebral and systemic oxymetry (rSO2) using near infrared spectroscopy (NIRS, Invos 5100; Somanet- ics Corporation, Troy, MI) will be performed on all patients with 4 optodes (right and left temporal area, arm and leg). Continuous rSO2 values will be stored on a hard disk with a 15 seconds update within intraoperative period and first 4 hours after the surgery. Desaturation phases (saturation decrease more than 20% of the basal value for more than 15 seconds) will be correlated to operative procedure or events. Postoperative adverse events will be collected. A correlation between desaturation and postoperative adverse events will be done with a multiple linear regression model.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing an hepatic resection or hepatic transplantation
* patients able to give consent with knowledge of french or english language.

Exclusion Criteria:

* age< 18 years
* patients with cerebral diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient undergoing hepatic surgery or liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
define the correlation coefficient between the number of systemic and/or cerebral desaturation phases and the number of postoperative adverse events | from the beginning of anesthesia till 4 hours after the end of the surgery

SECONDARY OUTCOMES:
define the prevalence of systemic and cerebral desaturation phases during hepatic surgery or transplantation | from the beginning of anesthesia till 4 hours after the end of the surgery
define the correlation coefficient between systemic and/or cerebral desaturation phases and the length of stay in intensive care unit | duration of intensive care stay, an expected average of 4 days
validate the equivalence of the systemic and cerebral oxymetry | from the beginning of anesthesia till 4 hours after the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Franck Vandenbroucke-Menu, MD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal; Réal Lapointe, MD-FRCS, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal; André Denault, MD PhD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada